CLINICAL TRIAL: NCT06287385
Title: An Exploratory Real-world Study to Explore the Effects of a Goat-milk Based Formula on Gut Health and Related Health Benefits in Healthy, Term-born Chinese Young Children
Brief Title: An Exploratory RWE Study Exploring Effects of a Goat Milk Based Young Child Formula on Health Benefits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NELN202212A
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2024-08

CONDITIONS: Healthy Children

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Formula fed (Experimental): Goat-milk Based Formula (Stage 3)
  Interventions: Dietary Supplement: Goat-milk Based Formula

INTERVENTIONS:
Dietary Supplement: Goat-milk Based Formula — Provided Goat-milk Based Formula for babies 1-2 years old

SUMMARY:
This is an exploratory real-world study designed to gain insight into the role of the product in terms of health benefits in toddlers, with the potential to generate hypotheses on key and other exploratory objectives.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 1-2 years of age
2. Healthy term infants, gestational ages 37~42 weeks
3. Birth weight within normal range for gestational age and sex (10th to 90th percentile of the Chinese Child Growth Chart);
4. Normal weight, height at screening (10th to 90th percentile of the Chinese Child Growth Chart)
5. Chinese population;
6. Subjects whose parents/guardians are intending to goat formula feed according to protocol during the study period;
7. Informed consent from one parent or legal representative;
8. Subjects whose parents/guardians are adults, have sufficient ability in Chinese to complete informed consent and other study documents;
9. Subjects whose parents/guardians are able to use smart phone with cameras; install and use a secure WeChat platform on the mobile phone during the study period; connect to the network through the mobile phone; take photos to record stool; complete questionnaires;
10. Subjects whose parents/guardians can be directly contacted by telephone or WeChat throughout the study.

Exclusion Criteria:

1. Probiotics or probiotics-supplemented products use within 4 weeks prior to enrolment;
2. Goat-milk based formula or fresh goat milk use within 4 weeks prior to enrolment;
3. Special infant formula use within 4 weeks prior to enrolment, including but not limited to hydrolysed infant formula, lactose-free infant formula and anti-reflux infant formula etc.;
4. Known allergy to milk products or soy product;
5. Medially diagnosed disorders requiring a special diet, including but not limited to reflux esophagitis, phenylketonuria etc;
6. Significant congenital abnormality or other health conditions that could affect the outcome measurements;
7. Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements;
8. Participation in any other studies involving investigational or marketed products concomitantly or within 4 weeks prior to entry into the study.

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Stool characteristics | before and 7, 14, 21 and 28 days after administration of the investigational product
  Stool characteristics assessed with BITSS

SECONDARY OUTCOMES:
Gastrointestinal symptoms | before and 7, 14, 21 and 28 days after administration of the investigational product
  Gastrointestinal symptoms assessed with Gastrointestinal Symptom Questionnaire
Quality of life of subjects | before and 28 days after administration of the investigational product
  Quality of life of subjects assessed with Pediatric Quality of Life Inventory (PedsQL)
Lifestyle-related immune indicators | before and 28 days after administration of the investigational product
  Lifestyle-related immunity status reported by parents or medically diagnosed (indicated in the subject's medical file)

OTHER OUTCOMES:
Safety assessment includes adverse events as reported spontaneously by parents or collected by investigators. | screening until 4 weeks after product intervention
  Safety assessment includes adverse events as reported spontaneously by parents or collected by investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Zailing Li, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No